CLINICAL TRIAL: NCT03699904
Title: A Randomised, Double-blind, Placebo-controlled Trial to Evaluate the Effect of Epstein-Barr Virus Suppression in Chronic Obstructive Pulmonary Disease (EViSCO).
Brief Title: Epstein-Barr Virus Suppression in Chronic Obstructive Pulmonary Disease (EViSCO): a Phase 2 Randomised Control Trial
Acronym: EViSCO
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: In light of the evolving Covid19 pandemic ongoing study recruitment was felt to pose an unacceptable risk to patient safety.
Sponsor: Belfast Health and Social Care Trust (Other)
Collaborators: Northern Ireland Clinical Trials Unit (Other); Queen's University, Belfast (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14143JK-AS
Record Dates: First submitted 2018-10-01; First posted 2018-10-09 (Actual); Last update posted 2020-09-30 (Actual); Status verified 2020-09

CONDITIONS: COPD; EBV
Keywords: COPD; EBV
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Valacyclovir

STUDY DESIGN:
Intervention Model Description: Parallel assignment.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This will be randomised, double-blind trial with matching placebo.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active arm (Experimental): Valaciclovir 1 gram orally three times daily for 8 weeks.
  Interventions: Drug: Valaciclovir
- Placebo arm (Placebo Comparator): Matching placebo capsules (containing Avicel blend). Two capsules three times daily for 8 weeks.
  Interventions: Drug: Placebo capsules (containing Avicel blend)

INTERVENTIONS:
Drug: Valaciclovir — Participants will self-administer Valaciclovir 1 gram three times daily for 8 weeks.
  Arms: Active arm
Drug: Placebo capsules (containing Avicel blend) — Participants will self-administer two matching placebo capsules (containing Avicel blend) three times daily for 8 weeks.
  Arms: Placebo arm

SUMMARY:
COPD is a major public health problem and will shortly become the third most common cause of global mortality. There are currently no treatments that can meaningfully alter the progression of COPD or the time to death. Consequently novel therapeutic strategies for COPD are urgently required. This will be a randomised, double-blind, placebo-controlled, trial of Epstein-Barr virus suppression in COPD. Participants will be randomised to receive valaciclovir 1 gram three times daily for 8 weeks or matching placebo. The study will measure EBV suppression using quantitative PCR. Secondary outcomes will include Lung function quality of life and drug tolerability. The exploratory analysis will evaluate biomarkers of airway inflammation within the sputum and blood.

DETAILED DESCRIPTION:
The study will evaluate the role of antiviral therapy in COPD. Previous research has demonstrated that Epstein-Barr virus (EBV) is more frequently identified in the airways of COPD sufferers when compared to unaffected smokers. It is not known whether suppression of EBV helps in COPD.

Hypothesis. The primary hypothesis is that treatment with valaciclovir is safe and will suppress Epstein-Barr virus in the sputum of patients with COPD.

Trial objectives. To conduct a randomised, double-blind, placebo-controlled, trial of Epstein-Barr virus suppression in COPD.

To evaluate the safety of valaciclovir (1 gram three times daily for 8 weeks) for the suppression of Epstein-Barr virus in COPD.

To study the biological effects of EBV suppression on airway and blood markers of inflammation in COPD.

The investigators will conduct a clinical trial to evaluate if a long established antiviral therapy (valaciclovir), routinely used to treat herpes zoster virus infection, can be used to suppress EBV shedding within the airways of COPD sufferers compared to placebo. The treatment will be randomised and blinded to both patients and investigators. The trial will recruit 88 participants who will undergo lung function testing, clinical assessment and provide blood and sputum samples at three separate hospital visits during an 8-week period (samples will be collected at 0, 4 & 8 weeks). A small subgroup of trial participants will undergo bronchoscopy on a voluntary basis to enable assessment of the airway cells before and after treatment. The study will take place in The Belfast Health and Social Care Trust. Patients who suffer from COPD (GOLD 2 & GOLD 3) and concurrent EBV infection will be eligible to participate in the study. If the treatment is effective this will lead to further research to determine whether antiviral therapy is effective in patients with COPD. The study will also provide new information about the mechanisms of how COPD develops and potentially identify new therapeutic targets.

Data management. The Northern Ireland Clinical Trials Unit (NICTU) will be responsible for data management during the conduct of the trial. Following electronic CRF submission data will be processed by NICTU as per CTU SOPs. All data will be anonymised. Data queries will be generated by site staff as required to clarify data or request missing information.

Data storage. All data and trial records will be stored by the CI in accordance with current regulatory requirements.

Sample size. A sample size of 31 subjects per group will have a 90% power at a two-tailed significance level of 0.05 to detect a difference in the exploratory efficacy outcome (EBV quantitative PCR).

Statistical analysis. Analyses will be on an intention-to-treat basis and all statistical tests will be at the 2-sided p-value of 0.05. Comparison between groups for the primary outcome measure SARs will be made using Fisher's exact test.

The exploratory efficacy outcome EBV shedding will initially be analyzed by chi-square test followed by logistic regression with adjustment for covariates if required. The comparison of continuous secondary/exploratory outcomes will be initially by t-tests followed by analysis of covariance if adjustment for covariates is required. Statistical diagnostic methods will be used to check for violations of the assumptions, and transformations will be performed where required.

Correlations between changes in the biological markers measured and physiological and clinical outcomes will be assessed by appropriate graphical and statistical methods including Pearson's (or Spearman's) correlation coefficient.

A single final analysis is planned at the end of the trial.

A detailed statistical analysis plan will be written before the statistical analysis commences.

ELIGIBILITY:
Inclusion Criteria:

1. Age over 18 years.
2. Clinical diagnosis of COPD as defined by the Global Initiative for Chronic Obstructive Lung Disease criteria (FEV1/FVC <70%) with GOLD 2 and GOLD 3 airflow obstruction (FEV1 30-80% predicted) with significant symptoms.
3. Presence of Epstein-Barr virus on sputum PCR analysis.

Exclusion Criteria:

1. Respiratory failure (defined as long-term oxygen therapy).
2. An acute exacerbation of COPD in the previous month (defined as an acute, sustained worsening of symptoms that is beyond normal day-to-day variations).
3. A diagnosis of asthma.
4. Patients with known hypersensitivity to valaciclovir or aciclovir.
5. Patients unable to swallow study drug capsules.
6. Established diffuse interstitial lung disease (e.g. Idiopathic Pulmonary Fibrosis).
7. Established diagnosis of symptomatic bronchiectasis.
8. Patients known to be pregnant or breastfeeding.
9. Patients with an estimated creatinine clearance less than 50ml/minute.
10. Known participation in investigational medicinal product trials within 30 days.
11. Patients who do not adequately understand verbal or written information.
12. Concomitant use of nephrotoxic medicinal products or medicines associated with altered renal tubular secretion. These include aminoglycosides, organoplatinum compounds, methotrexate, pentamidine, foscarnet, ciclosporin, tacrolimus,tenofovir, cimetidine and probenecid. As iodinated contrast used in radiological examinations can be nephrotoxicity patients with planned radiological contrast studies will be deferred for a reasonable time until after their contrast.
13. For the exploratory bronchoscopy sub-study patients will require adequate oxygen saturations, FEV1 >0.5 L and will not be performed while patients are taking aspirin or clopidogrel (BTS guidelines 2013).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2018-10-11 (Actual); Primary Completion 2020-05-07 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Incidence of Serious Adverse Reactions (SARs) | Up to 28 days after completion of the study drug
  The primary outcome measure will be drug safety of valaciclovir (1 gram three times daily for 8 weeks) as defined by the incidence of Serious Adverse Reactions (SARs).
EBV viral load | Change from baseline to 8 weeks.
  The primary efficacy outcome is suppression of Epstein-Barr virus in the sputum measured using quantitative PCR at baseline and 8 weeks.

SECONDARY OUTCOMES:
Forced expiratory volume in 1 second (FEV1) | Change from baseline to 8 weeks
  Lung function measured by spirometry, the principal component will be the change in FEV1 from baseline to week 8.
Drug tolerability as measured by the proportion of tablets self-administered. | 8 weeks
  Drug tolerability will be measured by total number of tablets self-administered as a proportion of total number of tablets supplied.

OTHER OUTCOMES:
COPD assessment test (CAT) score | Change from baseline to 8 weeks
  This instrument is a disease specific questionnaire that can quantify the impact of COPD on the patient's health. The CAT has a scoring range of 0-40. Higher scores indicate more severe impact of COPD.
EQ-5D-5L health status questionnaire | Change from baseline to 8 weeks
  The EQ-5D-5L is a standardised questionnaire designed to measure health status (quality of life) in patients. The EQ-5D-5L comprises five dimensions (mobility, self-care, usual activities, pain/discomfort and anxiety/depression). Each dimension may be scored from one to five enabling the description of 3125 different health states.

CONTACTS AND LOCATIONS:
Overall Officials: Joe Kidney, MB, MD, Principal Investigator — Belfast Health and Social Care Trust
Locations (1):
- Belfast Health and Social Care Trust, Belfast, Down, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Linden DA, Guo-Parke H, McKelvey MC, Einarsson GG, Lee AJ, Fairley DJ, Brown V, Lundy G, Campbell C, Logan D, McFarland M, Singh D, McAuley DF, Taggart CC, Kidney JC. Valaciclovir for Epstein-Barr Virus Suppression in Moderate-to-Severe COPD: A Randomized Double-Blind Placebo-Controlled Trial. Chest. 2023 Sep;164(3):625-636. doi: 10.1016/j.chest.2023.03.040. Epub 2023 Apr 1. PMID 37011709